CLINICAL TRIAL: NCT02294253
Title: Buprenorphine/Naloxone Stabilization and Induction Onto Injection Naltrexone: An Outpatient Detoxification for Opioid Dependence.
Brief Title: Buprenorphine/Naloxone Stabilization and Induction Onto Injection Naltrexone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Professor in Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6999
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Buprenorphine/naloxone stabilization (Experimental): Participants who have initially failed outpatient induction onto XR-NTX will receive buprenorphine/naloxone (BUP) on a weekly basis that they will take daily,
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — 30 day oral Buprenorphine/naloxone
  Other Names: Suboxone

SUMMARY:
The investigators will randomize 50 opioid-dependent participants who have initially failed outpatient induction onto XR-NTX; participants will receive buprenorphine/naloxone on a weekly basis for 30 days. Buprenorphine/naloxone will be dispensed weekly during the 30-day stabilization and twice weekly during taper phase, and all patients who successfully complete the detoxification will be offered induction onto XR-NTX. All participants will receive weekly therapy with a study psychiatrist. All participants will receive open-label medication. The primary outcome of this study will be percentage of patients successfully inducted onto XR-NTX. Secondary outcomes will be time to relapse, defined as opioid use or dropout.

DETAILED DESCRIPTION:
Buprenorphine induction/stabilization/taper: Buprenorphine induction will be conducted at our STARS clinic and according to current clinical guidelines. Participants who have initially failed outpatient induction onto XR-NTX will receive buprenorphine/naloxone (BUP) on a weekly basis that they will take daily, according to the following schedule: 8/2 mg (Days 1-10), 6/1.5 mg (Days 11-15), 4/1 mg (Days 16-20), 3.0/0.75 mg (Days 21-25), 2.0/0.5 mg (Days 26-30).

Participants will attend the clinic twice weekly and will be assessed for opioid and other substance use (urine toxicology and self-report), vital signs, opioid withdrawal symptoms, opioid cravings, and dose adjustments of buprenorphine will be made as needed by study physicians. If a dose reduction is needed, the stabilization and taper schedule will be adjusted to occur over 30 days.

Participants will be stabilized on, and tapered off, buprenorphine over a 4-week period.Reductions will occur in a graded fashion, with the stabilization dose reduced to 2 mg. This approach to buprenorphine taper is intended to resemble standard clinical practice, in which patients seeking transition off buprenorphine undergo a slow taper. A gradual taper over approximately 4 weeks has established precedent (Sigmon et al. 2013, Ling et al. 2009, Nielsen et al. 2013) as a well-tolerated taper strategy for transitioning off buprenorphine. The purpose is in part to provide a slow transition with minimal withdrawal symptoms. Participants will have at least two study visits a week during the buprenorphine taper, but may be seen more regularly at STARS if deemed clinically necessary.

Naltrexone induction procedure: Participants who successfully complete the taper must then complete a two-day washout (abstinence for opioids, buprenorphine). During this 48-hr period,participants will report to the STARS clinic daily for vital sign monitoring and to receive ancillary medications (clonidine, clonazepam, zolpidem, prochlorperazine) to alleviate withdrawal and discomfort as needed. After abstinence of >/=48 hours from the last buprenorphine dose, to allow for mu receptor availability, participants will begin the naltrexone induction,using a 4-day ascending taper of oral naltrexone (1, 3, 12, and 25 mg), followed by injection naltrexone . The administration of naltrexone will occur within a detoxification suite provided at STARS, consisting of a private room outfitted with two comfortable reclining lounge chairs for resting, adjustable lighting, and an entertainment system. Participants will be monitored by clinical staff at least every 1-2 hours with frequent vital signs checks and withdrawal assessments. A research psychiatrist or study physician will be present at all times to conduct frequent clinical assessments and provide adjuvant medications and naltrexone. Patients will be monitored on a daily basis (Monday to Friday) for up to 8 hours per day. Transportation home by car service will be provided at the end of the day for any patient deemed to have this clinical need.

On Day 1 of the naltrexone induction,participants are pre-treated with prochlorperazine 10 mg for nausea, followed be the first dose of naltrexone 1mg. Ascending doses of naltrexone will then be titrated upward slowly (3mg, 12mg, 25mg). Adjuvant medications will be available to patients and will include clonidine for myalgias, prochlorperazine for nausea, clonazepam to reduce anxiety and dysphoria, and trazodone or zolpidem for insomnia. Participants will be provided take-home doses of adjuvant medications in small doses and on a tapering schedule for one week post-administration of XR-NTX. Participants will be required to visit the clinic daily and remain there for at least 1 hour to permit close monitoring, with an option to stay as long as necessary to achieve relief of symptoms and medical stability prior to being discharged home.

Once 25 mg of naltrexone has been tolerated, the participant may receive 380 mg IM XR-NTX.

Additionally, for female participants, a urine pregnancy test will be obtained on the day of XR-NTX administration. Prior to administration of XR-NTX, participants who have been non-compliant with the oral naltrexone schedule, accompanied by lapses to opioid use, or in any case for which the challenge appears clinically indicated in the judgment of the study physician or research team, will receive a naloxone challenge prior to XR-NTX administration. Referrals to local treatment providers will be arranged for participants who successfully complete the study and request to continue XR-NTX maintenance

XR-NTX injections: XR-NTX will be administered once naltrexone 25 mg has been tolerated, as an intramuscular injection (380 mg) in one buttock by one of the research psychiatrists or research nurses of STARS, who are currently trained and administer XR-NTX in other protocols. Participants will be observed for at least 2 hours after the first injection. Participants will be offered a second injection at Week 5 (four weeks post-administration of the first injection), and a third injection at Week 9. Prior to receiving second and third injections at STARS, patients will either provide an opioid-negative urine or pass a naloxone challenge test.

At each STARS visit the patient meets with the research assistant to complete research ratings, including self-report of withdrawal, mood, and drug use. Blood samples are drawn according to the protocol for naltrexone serum levels and liver enzymes. The patient provides a urine sample under observation by a staff member at each visit. STARS is staffed by both male and female research assistants so that all urines can be appropriately monitored.

All participants will receive a weekly medication adherence-focused psychosocial intervention informed by relapse prevention strategies we previously developed in Behavioral Naltrexone Therapy and delivered by the study physician (Rothenberg, Sullivan et al. 2002). We have developed a relapse prevention approach which includes an emphasis on compliance with NTX. Participants will receive this therapy during weekly visits in outpatient Weeks 1-12 following induction onto XR-NTX.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60.
2. Meets DSM-IV criteria for current opiate dependence disorder of at least six months duration, supported by urine toxicology OR COWS score > or =6 OR Naloxone Challenge.
3. Voluntarily seeking treatment for opioid dependence.
4. In otherwise good health based on complete medical history and physical examination.
5. Able to give written informed consent.
6. Failed outpatient induction onto XR-NTX in Protocol #6374.

Exclusion Criteria:

1. Methadone maintenance treatment or regular use of illicit methadone (> 30 mg per week).
2. Maintenance on, or regular use of, buprenorphine or other long-acting opioid agonists.

3.) Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods. 4) Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with AST or ALT > 3 times normal, AIDS, unstable diabetes.

5) Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-5 Schizophrenia or any psychotic disorder, severe Major Depressive Disorder, or suicide risk or 1 or more suicide attempts within the past year.

6) Physiologically dependent on alcohol or sedative-hypnotics with impending withdrawal. Other substance use diagnoses are not exclusionary.

7) History of allergic or adverse reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.

8) Chronic organic mental disorder (e.g. AIDS dementia). 9) History of accidental drug overdose in the last 3 years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.

10) Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Evans, M.D., Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine/Naloxone Stabilization: Participants who have initially failedoutpatient induction onto XR-NTX will receive buprenorphine/naloxone (BUP) on a weekly basis that they will take daily,
  Buprenorphine/naloxone: 30 day oral Buprenorphine/naloxone
Period: Overall Study
Arm/Group | Buprenorphine/Naloxone Stabilization
Started | 30
Completed | 15
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine/Naloxone Stabilization
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Successful Induction Onto XR-NTX
Description: Proportion of participants inducted onto XR-NTX at the end of the 30-day buprenorphine/naloxone stabilization/taper.
Time Frame: One week after completing 30-day buprenorphone/naloxone stabilization/taper.
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone Stabilization
Number analyzed (Participants) | 30
Participants | 8

ADVERSE EVENTS:
Time Frame: AEs will be collected at each visit for the overall duration of the study which up to 3 months
Arm/Group | Buprenorphine/Naloxone Stabilization
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone Stabilization (N=30)
Priapism (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone Stabilization (N=30)
Insomnia (Psychiatric disorders) | 2 (2)
Decreased Appetite (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (3)
Decreased energy (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02294253/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02294253/SAP_001.pdf